CLINICAL TRIAL: NCT02330224
Title: Management of Hypertension and Multiple Risk Factors to Enhance Cardiovascular Health - A Cluster Randomized Pilot Trial in SingHealth Polyclinics, Singapore
Brief Title: Management of Hypertension and Multiple Risk Factors to Enhance Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke-NUS Graduate Medical School (Other)
Responsible Party: Principal Investigator, Professor Tazeen Jafar, Professor, Duke-NUS Graduate Medical School
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013/663/E
Record Dates: First submitted 2014-12-28; First posted 2015-01-01 (Estimated); Last update posted 2015-01-01 (Estimated); Status verified 2014-12

CONDITIONS: Hypertension; Cardiovascular Diseases
Keywords: Blood pressure; Lipids; Cardiovascular; Health services; Hypertension
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypertension Management Intervention (Experimental): Multifaceted hypertension management intervention
  Interventions: Other: Hypertension Management Intervention
- Usual Care (No Intervention): Control group

INTERVENTIONS:
Other: Hypertension Management Intervention — The multifaceted intervention consists of three main components:
  1. Structured treatment algorithm with fixed dose antihypertensives for high cardiovascular disease risk patients
  2. Motivational conversation by nurses and nurse practitioners for high risk patients at baseline
  3. Telephone based follow-up for all patients by nurses
  Arms: Hypertension Management Intervention

SUMMARY:
High blood pressure (BP) is a serious public health problem responsible for heart attack, stroke and kidney failure. One in four adults in Singapore has hypertension. We propose a pilot study in 2 polyclinics in Singapore, 1 deliver a structured multi-component intervention and another usual care. A total of 100 adults with uncontrolled high blood pressure will be followed for 3 months. The intervention includes 1) algorithm-driven antihypertensive treatment for all patients using fixed-dose combination and lipid lowering for high risk patients, 2) motivational conversation for high risk patients; and 3) telephone based follow-ups of all patients by a team of physician supervised nurse practitioners and nurses. The change in BP will be compared between intervention and control groups. The structured care including the above mentioned components is likely to be more effective than usual care in lowering BP levels of patients with uncontrolled high blood pressure. Such a program is also likely to be more cost effective in terms of money spent for improving quality of patients' life. The findings of the pilot will inform the design of a larger cluster randomized trial in eight polyclinics in Singapore. If the main study is successful, the findings will be informative for policymakers to roll out intervention in all polyclinics and primary care centers across Singapore, and other countries with similar healthcare infrastructure.

DETAILED DESCRIPTION:
1. Background:

   Cardiovascular diseases (CVD) are the leading cause of disability and death in Singapore, and consume substantial healthcare resources. Uncontrolled hypertension confers the highest attributable risk of CVD. About one in four adults suffer from hypertension in Singapore, 50% of them have uncontrolled blood pressure (BP), and management is especially sub-optimal among those with concomitant diabetes or dyslipidemia. Evidence suggests that well structured programs of care delivery are effective in lowering BP and preventing CVD. However, there is lack of empirical data on such strategies in Singapore.

   The findings of the pilot will inform the design of a larger cluster randomized trial in eight polyclinics in Singapore. If proven effective in the main study, the information will be valuable in convincing the policy-makers to upscale strategies for enhancing management of hypertension and cardiovascular health within the primary health infrastructure of Singapore, and possibly neighbouring Southeast Asian countries.
2. Aims:

   Specific aim 1: To explore logistics for delivery of provider training in intervention algorithm and motivational counselling while maintaining optimal efficiency of ongoing clinical work at the polyclinics.

   Specific aim 2: To establish recruitment of participants in the intervention and usual care groups, and uptake of each component of the multicomponent intervention.

   Specific aim 3: To establish mechanism for capture and retrieval of the relevant clinic visit data (physician and nurses records, pharmacy and laboratory including costs) at the polyclinic, and telephone follow-ups, hospitalization and related costs.

   Specific aim 4: To explore impact of intervention vs usual care on change in BP in the short term.

   Specific aim 5: Identify appropriate methods for capturing potential adverse events and safety endpoints related to intervention.
3. Study Design: It is a non-randomized community intervention trial designed to test feasibility of structured multi-component intervention in polyclinic setting.
4. Setting: The study involves two polyclinics in Singapore. One delivers intervention and one delivers usual care.
5. Study population: The polyclinics have a system in place such that all patients with hypertension get a "panel" of fasting blood and urine tests at subsidized cost at the time of initial diagnosis and then annually. The individuals visiting polyclinic for their initial (or annual) panel of laboratory tests marked as "hypertension panel" will be screened for eligibility and recruited if eligible. One hundred patients (50 per polyclinic) will be recruited and followed for 3 months.
6. Intervention: Orientation training sessions will be organized for all physicians, nurse practitioners (NP) and nurses in the polyclinic assigned the intervention which is comprised of 3 components

   1. Structured treatment algorithm with fixed dose antihypertensives for high risk patients: The training curriculum including treatment algorithm has been prepared by a team of nephrologists, cardiologists and pharmacologists in consultation with primary care physicians and Clinical Cardiovascular Work Group, using the case method, aiming for global cardiovascular risk reduction.
   2. Motivational conversation by NPs and nurses for high risk patients at baseline: Separate training sessions will be conducted for NP and nurses. NP and nurses will receive training on motivational conversation techniques and communication strategies from a trainer skilled in communication in health care. These nurse and nurse practitioners will provide motivational conversation sessions to high CVD risk patients at baseline.
   3. Structured follow-up over telephone and in Clinics: NPs and nurses in intervention polyclinic will be proactive in follow-up of their patients for self-monitoring of BP and providing advice for adherence to treatment every 4 weeks for the duration of the project (3 months). A communication checklist for the follow-up will be incorporated to the existing follow-up system. Information on adverse events will be obtained and action plan will be communicated with patients (discontinue the suspected drug and arrange visit to clinic, as appropriate).
7. Usual Care: The health providers in the polyclinic with usual care will continue their existing practices.
8. Outcomes assessment: Final outcome assessment will take place three months after baseline. The outcomes assessors will also call the patients over telephone for outcomes assessment at week 6 after baseline. Information on self-monitoring of BP, recommended life style change, self-care, and medication use (including herbal and traditional Chinese) will be collected.

   The outcome assessors will also extract process outcomes measures from the general practitioner (GP) and nurses' notes. These will include number and duration of contact with the patient (whether in person or by phone), changes in prescribed medication and dose, and reporting of any adverse events from medications.
9. Sample size calculation: Sample size was calculated using Stata version 12. A sample size of 90 (45 in each group) achieves 80% power to detect 5 mmHg difference in systolic BP change from baseline to end of follow-up in intervention group compared to usual care group, with an estimated standard deviation (SD) of 9.5, significance level of 0.05 using a two-sided two-sample t-test. Assuming that there could be 10% drop out rate, we plan to take the total sample size of 100 subjects. At least 152 eligible subjects (72 in each group) would be necessary to attain at least 66% recruitment rate.

ELIGIBILITY:
Inclusion Criteria:

* 40 years or older
* Singapore citizen and Permanent Resident
* Individuals visiting the recruiting polyclinic at least twice during the last 1 year
* Individuals with with previously diagnosed hypertension and uncontrolled blood pressure (Systolic BP 140 mmHg and above and diastolic BP 90 mmHg)

Exclusion Criteria:

* Individuals with active systemic illness including fever
* Individuals with recent hospitalization (i.e. during last 4 months),
* Individuals with clinically unstable heart failure (i.e. Ejection fraction <20% or complaint of shortness of breath at rest)
* Individuals with advanced kidney disease (i.e. estimated Chronic kidney disease (CKD) -Epi glomerular filtration rate <40 ml/min/1.73m2 or nephrotic range proteinuria (i.e. 3g/d or more))
* Individuals with known advanced liver disease (i.e. Child-Pugh Stage C)
* Individuals with pregnancy
* Individuals with any other major debilitating disease or
* Individuals with mental illness that precludes validity of informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in Systolic Blood Pressure from baseline to final follow-up at 3 months | Baseline, month 3

SECONDARY OUTCOMES:
Proportion of planned orientation sessions delivered | Baseline
  Orientation training session for treatment algorithm and motivational counseling will be organized in multiple lunch-time sessions. The number of orientation sessions planned will be denominator and the number of sessions successfully delivered will be numerator. Target is 100%.
Percent uptake of motivational interviewing sessions | 3 months
Percent of data (laboratory and medication) retrieved from the polyclinic electronic database | At month 3
  The total number of participants received the laboratory tests and prescribed medications will be denominators and the number of participants whose data are successfully retrieved from electronic database will be numerator. Target is 98% of data retrieved.
Proportion of blood pressure readings obtained at final follow-up | At month 3
  Total number of participants enrolled will be denominator. Number of participants whose blood pressure readings are successfully obtained at final visit (3 months from baseline) will be numerator. Target is 80%.
Proportion of participants recruited | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tazeen H Jafar, MD, MPH, Principal Investigator — Duke-NUS Graduate Medical School; Ngiap Chuan Tan, MBBS, Principal Investigator — SingHealth Polyclinics, Research
Locations (2):
- Singapore (2):
  - SingHealth Polyclinics, Geylang, Singapore
  - SingHealth Polyclinics, Tampines, Singapore

REFERENCES:
- [Derived] Jafar TH, Tan NC, Allen JC, Pradhan SS, Goh P, Tavajoh S, Keng FM, Chan J. Management of hypertension and multiple risk factors to enhance cardiovascular health - a feasibility study in Singapore polyclinics. BMC Health Serv Res. 2016 Jul 8;16:229. doi: 10.1186/s12913-016-1491-6. PMID 27391818